CLINICAL TRIAL: NCT00269399
Title: A Double-Blind, Randomized, Controlled Trial of Rifaximin Compared to Vancomycin for the Treatment of Clostridium Difficile-Associated Diarrhea (CDAD)
Brief Title: A Trial to Compare Xifaxan to Vancomycin for the Treatment of Clostridium Difficile-Associated Diarrhea (CDAD)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RFCL3001
Record Dates: First submitted 2005-12-22; First posted 2005-12-23 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-09

CONDITIONS: Clostridium Infections; Diarrhea
Keywords: Clostridium difficile-associated Diarrhea (CDAD); CDAD; C diff
MeSH Terms: conditions — Clostridium Infections; Diarrhea | interventions — Rifaximin; Vancomycin

ARMS (2):
- Rifaximin Treatment Arm (Experimental): rifaximin 400mg taken 3 times a day
  Interventions: Drug: Rifaximin (Xifaxan)
- Vancomycin Comparator Arm (Active Comparator): vancomycin 125mg taken 4 times a day
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Rifaximin (Xifaxan)
  Arms: Rifaximin Treatment Arm
Drug: Vancomycin
  Arms: Vancomycin Comparator Arm

SUMMARY:
The purpose of this study is to assess the treatment and safety of a 10-day course of rifaximin (Xifaxan) as compared to vancomycin for treatment of Clostridium difficile-associated diarrhea (CDAD).

DETAILED DESCRIPTION:
Clostridium difficile is a bacterium that proliferates when normal colonic flora have been altered, most commonly due to antibiotic use. Clostridium difficile is non-invasive and localized to the lumen of the colon. Once established, it produces 2 potent toxins, A and B. The principal reservoir for Clostridium difficile is the hospital environment, with the risk of acquiring Clostridium difficile increasing in direct proportion to the length of hospital stay.

Patients with CDAD typically present with profuse watery or mucoid diarrhea and cramping abdominal pain. Additional symptoms include fever, nausea, anorexia, malaise, and bloody stool. More severe cases may be complicated by dehydration, electrolyte disturbances, ileus, and peritonitis. Systemic manifestations may include prerenal azotemia, sepsis syndrome, and toxic colitis. White blood cell counts (WBCs) also may be markedly elevated with a shift to immature forms. Extreme presentation of fulminant colitis may require a colectomy and even result in death. Symptoms of CDAD may begin a few days after initiation of antibiotic therapy or up to 8 weeks after its discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Subject is 18 years of age or older, has acute diarrhea and at least 1 other sign of enteric infection present, such as fever, nausea/loss of appetite, vomiting, severe abdominal pain or discomfort.
* Subject has a positive Clostridium difficile stool toxin assay at screening

Exclusion Criteria:

* Subject has had a previous episode of clinically diagnosed Clostridium difficile within the past 6 months.
* Subject has chronic diseases associated with diarrhea (e.g., inflammatory bowel disease or diarrhea predominant irritable bowel syndrome [DIBS])
* Subject has had any therapy with any agent administered for the treatment of Clostridium difficile prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 237 (Actual)
Dates: Start 2005-12; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (63):
- United States (63):
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - Inland Empire Digestive & Liver Diseases, Redlands, California
  - Gastroenterology of the Rockies, Longmont, Colorado
  - Connecticut Gastroenterology Institute, Bristol, Connecticut
  - The George Washington University Medical Center, Washington D.C., District of Columbia
  - Halifax Medical Center, Daytona Beach, Florida
  - Advanced Medical Research Center, Port Orange, Florida
  - Webster Surgical Center LLC, Tallahassee, Florida
  - Digestive Healthcare of Georgia, Atlanta, Georgia
  - Southeast Regional Research Group, Columbus, Georgia
  - Sky Blue, M.D., Boise, Idaho
  - Howard Brown Health Center, Chicago, Illinois
  - The University of Chicago, Chicago, Illinois
  - Gastroenterology, Ltd., Peoria, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Clinic Association NCW5, Urbana, Illinois
  - Iowa Digestive Disease Center, PC, Des Moines, Iowa
  - GI Specialists, Olathe, Kansas
  - Gastrointestinal Associates, Overland Park, Kansas
  - Kansas Medical Clinic, Topeka, Kansas
  - Baltimore VA Medical Center, Baltimore, Maryland
  - University of Maryland, Baltimore, Maryland
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Center for Clinical Research at Washington County Hospital, Hagerstown, Maryland
  - Shah Associates, Prince Frederick, Maryland
  - Henry Ford Hospital, Detroit, Michigan
  - Arnold Markowitz, MD, PC, Keego Harbor, Michigan
  - Newland Medical Association, Southfield, Michigan
  - St. Mary's/Duluth Clinic Health System, Duluth, Minnesota
  - Minneapolis VAMC, Minneapolis, Minnesota
  - Infectious Disease - Minneapolis Ltd., Minneapolis, Minnesota
  - Mayo Clinic Rochester, Rochester, Minnesota
  - Digestive Health Specialists, PA, Tupelo, Mississippi
  - Deaconess Billings Clinic Research, Billings, Montana
  - Infectious Diseases Associates, PC, Omaha, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Drs. Scherl, Chessler, Zingler, Spinnel and Meininger, Fort Lee, New Jersey
  - Marlboro Gastroenterology PC, Manalapan, New Jersey
  - St. Michael's Medical Center, Newark, New Jersey
  - Institute for Clinical Research (ICR) at Holy Name Hospital, Teaneck, New Jersey
  - The Gastroenterology Group of South Jersey, Vineland, New Jersey
  - Brookdale University Hospital and Medical Center, Brooklyn, New York
  - AMS Clinical Research, Elmira, New York
  - North Shore Hepatology, Manhasset, New York
  - Weill Medical College, New York, New York
  - University of Rochester School of Medicine, Rochester, New York
  - New York Medical College/Westchester Medical Center, Valhalla, New York
  - East Carolina Gastroenterology, PA, Jacksonville, North Carolina
  - Southern Gastroenterology Associates, New Bern, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Regional Infectious Diseases - Infusion Center, Lima, Ohio
  - Lima Memorial Health System, Lima, Ohio
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - RPS Infectious Diseases, West Reading, Pennsylvania
  - University Gastroenterology, Providence, Rhode Island
  - Digestive Disease Associates of Dallas, Dallas, Texas
  - Michael E. DeBakey VA Medical Center, Houston, Texas
  - University of Texas Health Sciences Center, Houston, Texas
  - Infectious Disease Associates of Central Virginia, Lynchburg, Virginia
  - North Pacific Clinical Research, Redmond, Washington
  - Associated Physicians, LLP, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Rifaximin Treatment Arm: rifaximin 400mg taken 3 times a day
  Rifaximin (Xifaxan)
Period: Overall Study
Arm/Group | Rifaximin Treatment Arm | Vancomycin Comparator Arm
Started | 119 | 118
Completed | 78 | 91
Not Completed | 41 | 27
Not completed — Lack of Efficacy | 27 | 10
Not completed — Adverse Event | 10 | 4
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Negative Lab Result for C. difficile | 2 | 3
Not completed — Other | 0 | 4
Not completed — Development of exclusion criteria | 0 | 1

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-Treat (MITT) population included all randomized subjects who had acute diarrhea and with a positive C. difficile stool toxin assay within ± 48 hours of screening and received at least one dose of study drug.
Groups:
- Vancomycin Comparator Arm: vancomycin 125mg taken 4 times a day
  Vancomycing
- Total: Total of all reporting groups
Arm/Group | Rifaximin Treatment Arm | Vancomycin Comparator Arm | Total
Number analyzed (Participants) | 117 | 115 | 232
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.9 (16.22) | 60.0 (18.08) | 59.5 (17.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 67 | 141
  Male | 43 | 48 | 91
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 12 | 26
  White | 103 | 102 | 205
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Achieving Clinical Success, Where Clinical Success is Defined as Resolution or Improvement of Baseline Signs and Symptoms i.e., Abdominal Pain, Fever, Diarrhea.
Description: Resolution or improvement of baseline signs and symptoms was assessed as
  * Absence of severe abdominal pain for 2 consecutive days at the test of cure (TOC) Visit (Day 14 +/-1);
  * Absence of fever (< 38°C/100.4°F) for 2 consecutive days at the TOC Visit; and
  * 3 unformed (loose or watery) stools per day for at least 48 hours that was sustained through the TOC Visit.
Time Frame: 14 days
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Groups:
- Vancomycin Comparator Arm: vancomycin 125mg taken 4 times a day
  Vancomycin
Arm/Group | Rifaximin Treatment Arm | Vancomycin Comparator Arm
Number analyzed (Participants) | 117 | 115
Participants | 67 | 73

2. Secondary Outcome: Proportion of Participants Recurrence-free of Clostridium Difficile-associated Diarrhea (CDAD), After Achieving Clinical Success
Description: Recurrence of CDAD was defined as diarrhea and a positive Clostridium difficile stool toxin assay that occurs after initial clinical success.
Time Frame: 42 days
Population: Participants included in this analysis were restricted to those who experienced initial clinical success at the TOC Visit following the 10-day Treatment Phase.
Measure: Count of Participants; unit: Participants
Arm/Group | Rifaximin Treatment Arm | Vancomycin Comparator Arm
Number analyzed (Participants) | 67 | 73
Participants | 61 | 63

ADVERSE EVENTS:
Time Frame: 42 days
Description: For safety analyses participants are counted based on the treatments received rather than randomization assignment; 120 participants in the rifaximin group and 116 participants in the vancomycin group. Two (2) participants in the vancomycin group are handled differently than as randomized, including 1 participant who did not receive study drug (so excluded from the safety population) and 1 participant counted in the rifaximin group for safety since the subject actually received rifaximin.
Arm/Group | Rifaximin Treatment Arm | Vancomycin Comparator Arm
Serious Adverse Events (participants affected / at risk) | 28/120 | 14/116
Other Adverse Events (participants affected / at risk) | 6/120 | 2/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rifaximin Treatment Arm (N=120) | Vancomycin Comparator Arm (N=116)
Anemia (Blood and lymphatic system disorders) | 1 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 4 | 0
Diarrhea (Gastrointestinal disorders) | 3 | 3
Pyrexia (General disorders) | 1 | 1
Clostridial infection (Infections and infestations) | 2 | 1
Clostridium colitis (Infections and infestations) | 2 | 0
Pneumonia (Infections and infestations) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 3 | 4
Mental status changes (Psychiatric disorders) | 0 | 2
Renal failure acute (Renal and urinary disorders) | 3 | 2
Hypotension (Vascular disorders) | 3 | 2
Anemia hemolytic autoimmune (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1
Colitis ulcerative (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Umbilical hernia (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Asymptomatic bacteriuria (Infections and infestations) | 1 | 0
Bacteremia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Klebsiella sepsis (Infections and infestations) | 1 | 0
Pseudomonas infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 1 | 0
Collapse of lung (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 1
Blood creatinine increased (Investigations) | 1 | 0
Blood urea increased (Investigations) | 1 | 0
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung meoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
Chromic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hydopneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rifaximin Treatment Arm (N=120) | Vancomycin Comparator Arm (N=116)
Insomnia (Psychiatric disorders) | 6 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact sponsor for details.